CLINICAL TRIAL: NCT01323725
Title: The Effectiveness of Team-based Financial Incentives for Increasing Long-term Smoking Cessation
Brief Title: Team-based Financial Incentives for Smoking Cessation
Acronym: StPaulKorea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St.Paul's Hospital, Korea (Other)
Responsible Party: Principal Investigator, Sang Haak Lee, Professor, St.Paul's Hospital, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: StPaulKorea
Record Dates: First submitted 2011-03-25; First posted 2011-03-28 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Tobacco Use Disorder
Keywords: Team-based financial incentives; Smoking cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Team-based financial incentives (Experimental): Team-based financial incentives
  Interventions: Behavioral: Team-based financial incentives

INTERVENTIONS:
Behavioral: Team-based financial incentives — Team-based financial incentives for smoking cessation at 6 month post-quit date.

SUMMARY:
The purpose of this study is to identify the effectiveness of team-base financial incentives for increasing long-term smoking cessation among employees at St. Paul's Hospital, Korea.

DETAILED DESCRIPTION:
About 70% of smokers report that they want to quit, but annually 2 to 3% of smokers succeed. Smoking-cessation programs and pharmacologic therapies have been proven effective in helping smokers quit, but only a few smokers are enrolled in those programs.

Financial incentives may contribute to reinforce smoking cessation among workers through the following pathways: (1) increasing the number of tobacco users who participate in cessation effort; (2) increasing the number of tobacco user who initiate an attempt to quit; and (3) increasing the number of tobacco users who sustain a successful quit effort. Moreover, there is a number of advantages to offering smoking cessation support in the workplace, including the accessibility of the target population, the availability of occupational health support and the potential for peer pressure and peer support. In addition, team-based approach for smoking cessation could likely make use of new or existing cessation support resources offered within the workplace.

This study is a clinical trial of team-based financial incentives for smoking cessation among a sample of 60 smokers, who are health care workers from St. Paul's Hospital in Korea. Smokers will be given a usual care (counseling, education and coverage of prescription drugs) plus a package of financial incentives for self-reported and biochemically validated smoking cessation (urine or saliva cotinine). All incentives will be provided to each team at 6 months post-quit date.

ELIGIBILITY:
Inclusion Criteria:

* Employees of St. Paul's Hospital at work sites in Korea
* Current smoker who report having smoked at least 5 cigarettes per day for the prior 12 months
* Age 18 or older

Exclusion Criteria:

* Age 17 or younger
* Unwilling to quit smoking
* Smoker who does not want to be enrolled in this trial
* Planning to leave St. Paul's hospital within the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Smoking Cessation Rate | 6 months
  Self-reported and biochemically validated smoking cessation rate at 6 months post-quit date

SECONDARY OUTCOMES:
Smoking Cessation Rate | 3, 9, 12 months
  Self-reported and biochemically validated smoking cessation rate at 3, 9, 12 months post-quit date

CONTACTS AND LOCATIONS:
Overall Officials: Sang Haak Lee, MD, Principal Investigator — St. Paul's Hospital
Locations (1):
- St.Paul's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes